CLINICAL TRIAL: NCT04610281
Title: Pilot Study on the Care for Children With Moderate to Severe Agitation, With or Without the Use of a Semi-supervised Support Solution
Brief Title: The Inner Garden and Care for Children With Moderate to Severe Agitation
Acronym: ESSAIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Collaborators: Ullo World (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/P08/360
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-02

CONDITIONS: Child Behavior Disorders
MeSH Terms: conditions — Child Behavior Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Wards without the "Inner Garden" biofeedback tool
- Inner Garden (Experimental): Wards with the "Inner Garden" biofeedback tool
  Interventions: Device: Inner Garden

INTERVENTIONS:
Device: Inner Garden — Care actions adapted to the intensity of the states of agitation (The child can be removed from the group while remaining in the same room on a chair with a caregiver. If the problems are too serious, the child can be accompanied to a "soothing" room where the carer will take care of him/her individually. In units equipped with Inner Garden, the child can use it under semi- supervision of nurses.)
  Arms: Inner Garden

SUMMARY:
The objective is to compare the care including the solution of ambient sensory biofeedback "Inner Garden", compared to the care without this solution, on the regulation of behavioral disorders during a crisis requiring to take the child out of group care. The nursing support with the "Inner Garden" tool in three care units will be compared with the practice in six other units not equipped with this tool.

DETAILED DESCRIPTION:
Psychiatric illnesses affect more than one person in five each year. In France, the majority of disorders among minors under the care of child psychiatry in full or part-time hospitalization are disorders of psychological development (32%) and behavioural and emotional disorders (24.6%). Hospitalisation is reserved for the most complex acute crisis situations, as well as for children who need to be cared for by a multidisciplinary team several times a week to support their psychological development. In our study, the investigators focus on one of the clinical manifestations regularly present: the state of agitation when its intensity is moderate to severe. "The state of agitation is defined as a psychic, motor and relational behavioural disorder that leads to a reaction of intolerance on the part of people in the entourage". The care teams will then implement care actions that will be a graduated response adapted to the intensity of these states of agitation. In addition to the support provided by a caregiver, the investigators propose to use the "Inner Garden" system developed in 2014 at the laboratory of National Institute for Research in Digital Science and Technology in Bordeaux. It is an interactive Zen garden allowing to present feedback (topographical, physiological) under different sensory modalities.

ELIGIBILITY:
Inclusion Criteria:

* Taken care in Children's Hospitalization Unit of Child Psychiatry Department,
* Parent affiliated or beneficiary of social security,
* Information to the child and the legal representative(s) and signed consent by the legal representative(s).

Exclusion Criteria:

* Refusal to participate on the part of the child and/or legal representative(s).

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nordine Benmabrouk, RN, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis; Brigitte Laurent, PhD, Study Director — Ullo World
Locations (1):
- Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available with publication. Keyword are Child Behavior, Psychomotor Agitation, Psychiatric Nursing, Child Day Care Center, Tool Use Behavior, Emotional Regulation.
  The available version will be the locked database. The database will be made available by the study director upon request up to 15 years after publication.
  Medical Subject Headings (MESH) terms will be used to describe clinical data. Methodology for will be provided in the publication.
  International standard unit will be used.
Time Frame: Data will be made available with publication (expected at the end of 2021 or beginning of 2022) and up to 15 years after the end of the study.
Access Criteria: The database will be made available by the study director upon request

REFERENCES:
- [Background] Domon-Archambault V, Terradas MM, Drieu D, De Fleurian A, Achim J, Poulain S, Jerrar-Oulidi J. Mentalization-Based Training Program for Child Care Workers in Residential Settings. J Child Adolesc Trauma. 2019 Jun 21;13(2):239-248. doi: 10.1007/s40653-019-00269-x. eCollection 2020 Jun. PMID 32549935
- [Background] Niquille M, Gremion C, Welker S, Damsa C. [Agitation in prehospital setting: view of emergency physicians]. Rev Med Suisse. 2007 Aug 15;3(121):1839-46. French. PMID 17892148
- [Background] Tereno S, Soares I, Martins C, Celani M, Sampaio D. Attachment styles, memories of parental rearing and therapeutic bond: a study with eating disordered patients, their parents and therapists. Eur Eat Disord Rev. 2008 Jan;16(1):49-58. doi: 10.1002/erv.801. PMID 17879224
- [Background] Lewis GF, Hourani L, Tueller S, Kizakevich P, Bryant S, Weimer B, Strange L. Relaxation training assisted by heart rate variability biofeedback: Implication for a military predeployment stress inoculation protocol. Psychophysiology. 2015 Sep;52(9):1167-74. doi: 10.1111/psyp.12455. Epub 2015 Jun 11. PMID 26095854
- [Background] Zeman J, Shipman K, Suveg C. Anger and sadness regulation: predictions to internalizing and externalizing symptoms in children. J Clin Child Adolesc Psychol. 2002 Sep;31(3):393-8. doi: 10.1207/S15374424JCCP3103_11. PMID 12149977
- [Background] Chicchi Giglioli IA, Pallavicini F, Pedroli E, Serino S, Riva G. Augmented Reality: A Brand New Challenge for the Assessment and Treatment of Psychological Disorders. Comput Math Methods Med. 2015;2015:862942. doi: 10.1155/2015/862942. Epub 2015 Aug 3. PMID 26339283
- [Background] Baus O, Bouchard S. Moving from virtual reality exposure-based therapy to augmented reality exposure-based therapy: a review. Front Hum Neurosci. 2014 Mar 4;8:112. doi: 10.3389/fnhum.2014.00112. eCollection 2014. PMID 24624073
- [Background] Gold G, Fazio L, Stolz JH, Herrman FR, Gattelet P, Zekry D. [Assessment of behavior in non-psychiatric settings: use of a simple and reliable method]. Rev Med Suisse. 2012 Nov 7;8(361):2119-21. French. PMID 23173347
- [Background] Kay SR, Wolkenfeld F, Murrill LM. Profiles of aggression among psychiatric patients. I. Nature and prevalence. J Nerv Ment Dis. 1988 Sep;176(9):539-46. doi: 10.1097/00005053-198809000-00007. PMID 3418327

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Inner Garden
Started | 30 | 33
Completed | 29 | 29
Not Completed | 1 | 4
Not completed — Improvement in their condition no longer justifies care in the Children's Hospital Unit | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Inner Garden | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 33 | 63
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.9 (1.8) | 7.2 (1.7) | 7.1 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 25 | 27 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 30 | 33 | 63
Home [Count of Participants; unit: Participants]
  Institution | 0 | 2 | 2
  Foster care | 3 | 6 | 9
  Family home | 27 | 25 | 52
Enrolled in school [Count of Participants; unit: Participants]
  Yes | 29 | 31 | 60
  No | 1 | 2 | 3
Reason for hospitalisation [Count of Participants; unit: Participants]
  Developmental disorders | 15 | 14 | 29
  Conduct and/or emotional disorders | 3 | 9 | 12
  Other (mental retardation, hyperkinetic, social, adjustment disorders, congenital malformations) | 6 | 6 | 12
  Observation for suspected psychiatric illness, unspecified | 6 | 4 | 10
Number of years of inpatient care for children [Mean (Standard Deviation); unit: years] | 2.8 (1.4) | 2.4 (1.3) | 2.6 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Crises
Description: Agitation crises of moderate to severe intensity, which did not allow the child to reintegrate the group of care during the sessions
  A mild state of agitation does not require the child to be removed from the group and from the common place of care; A moderate agitation requires removal of the child from the group but not from the common place of care; In case of serious agitation, the child must be removed from the group and from the common care area to a "calming" room where the caregiver will take care of him/her individually.
Time Frame: 8 months after inclusion
Measure: Number; unit: crises
Arm/Group | Control | Inner Garden
Number analyzed (Participants) | 30 | 33
crises | 97 | 35

2. Secondary Outcome: Score at the Emotion Regulation Checklist
Description: The ERC items assess affective stability, intensity, valence, flexibility, and situational appropriateness of children between the ages of 6 to 12 years.
  Items are rated by a parent on a 4-point scale (1=never, 2=sometimes, 3=often, 4=almost always) and are weighted both negatively and positively.
  The ERC is comprised of two scales: emotion regulation (10 items) and emotional lability/negativity (14 items).
  The former scale assesses expression of emotions, empathy, and emotional self-awareness, with higher scores indicating greater adaptive regulatory processes (range 10-40).
  The latter scale assesses lack of flexibility, anger dysregulation, and mood lability, with higher scores indicating greater emotion dysregulation (range 14-56).
  The Composite emotional regulation score is the sum of the emotion regulation score and the inverted emotional lability score with higher scores indicating greater adaptive regulatory processes (range 24-96).
Time Frame: 4 months after inclusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Inner Garden
Number analyzed (Participants) | 30 | 33
score on a scale
  Emotional regulation score | 21.8 (6.7) | 21.7 (3.8)
  Emotional Lability/Negativity score | 33.1 (10.5) | 34.9 (8.5)
  Composite emotional regulation score | 54.9 (11.6) | 56.6 (9.0)

3. Secondary Outcome: Score at the Emotion Regulation Checklist
Description: as for outcome 2
Time Frame: 8 months after inclusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Inner Garden
Number analyzed (Participants) | 29 | 29
score on a scale
  Emotional regulation score | 21.6 (4.2) | 22.5 (3.7)
  Emotional Lability/Negativity score | 32.0 (7.5) | 34.5 (7.6)
  Composite emotional regulation score | 53.6 (7.4) | 56.7 (7.3)

4. Secondary Outcome: Number of Child for Which Assault or Violence Against Health Care Professionals Was Reported
Description: Assault or violence against health professional with a statement in the dedicated application.
  In cases of severe agitation, the child's hetero-aggressive actions may injure the caregiver.
Time Frame: 9 months after inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Inner Garden
Number analyzed (Participants) | 30 | 33
Participants
  Assault or violence against health professional | 2 | 1
  No assault or violence against health professional | 28 | 32

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Control | Inner Garden
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 0/30 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT04610281/Prot_SAP_000.pdf